CLINICAL TRIAL: NCT03055741
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IIb, Clinical Study to Evaluate the Safety and Efficacy of DHP1401 in Patients With Mild-moderate Alzheimer's Disease Treated With Donepezil(DRAMA)
Brief Title: Study of DHP1401 in Patients With Mild-moderate Alzheimer's Disease Treated With Donepezil(DRAMA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1401CS-2
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Mild-moderate Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): donepezil: 5mg or 10mg is orally administrated once a day for 24 weeks
  DHP1401: Total 500mg is orally administrated in two divided doses a day for 24 weeks
  Interventions: Drug: Donepezil; Drug: DHP1401
- Group 2 (Experimental): donepezil: 5mg or 10mg is orally administrated once a day for 24 weeks
  DHP1401: Total 1,000mg is orally administrated in two divided doses a day for 24 weeks
  Interventions: Drug: Donepezil; Drug: DHP1401
- Group 3 (Placebo Comparator): donepezil: 5mg or 10mg is orally administrated once a day for 24 weeks
  DHP1401: Placebo is orally administrated in two divided doses a day for 24 weeks
  Interventions: Drug: Donepezil; Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — 5mg or 10mg, once a day, 24 weeks
  Other Names: Aricept®
Drug: DHP1401 — Total 500mg or 1,000mg was administrated in two divided doses a day for 24 weeks
  Other Names: DHP1401 500mg or 1,000mg
  Arms: Group 1; Group 2
Drug: Placebo — Placebo was administrated in two divided dosed a day for 24 weeks
  Other Names: DHP1401 placebo
  Arms: Group 3

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of DHP1401 in patients with mild-moderate Alzheimer's disease treated with donepezil

ELIGIBILITY:
Inclusion Criteria:

1. ≥55 and ≤85 years of age
2. Patient who was diagnosed mild to moderate Alzheimer's disease by National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association(NINCDS-ADRDA) or National Institute on Aging-Alzheimer's Association(NIAAA)
3. Korean Mini-Mental State Examination(K-MMSE) score 15 to 26
4. Patient who maintained on donepezil without dose escalation or reduction for at least during 3 months before screening (visit 1)
5. Clinical Dementia Rating(CDR) score 0.5 to 2.0 at screening (visit 1)
6. Written informed consent voluntarily
7. Patient who has a relative/caregiver who support the information of patient's status
8. Patient who are deemed adequate to participate in the clinical trial by the investigator
9. Infertility or patients and his/her spouse consent with contraception during the study period

Exclusion Criteria:

1. A diagnosis of vascular dementia or dementia by other cause according to the criteria of the NINCDS-ADRDA
2. Structural brain abnormality or impairment
3. Schizophrenia, depressive disorder and bipolar disorder
4. Any neurological disease except Alzheimer' disease (ex. Parkinson's disease, Huntington's disease, brain tumor, normal-pressure hydrocephalus, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, epilepsy, delusion and head injury required hospitalization)
5. History of any cancer within previous 5 years
6. History of stroke within previous 2 years
7. Heart failure required medication or interventional treatment including myocardial infarction, valvular heart disease, arrhythmia within previous 1 year
8. Uncontrollable diabetes
9. Uncontrollable hypertension
10. Abnormal liver or kidney function
11. Patient with significant clinical meaning to affect cognitive function
12. Patient who participated in other clinical trial within previous 3 months or has a plan to participate in other clinical trial during study period
13. History of abuse of a drug or alcohol within previous 2 years
14. Patient who has administrated other acetylcholinesterase inhibitors except donepezil within previous 4 weeks
15. Patient who are deemed inadequate to participate in the clinical trial by the investigator(ex. a illiteracy, etc.)
16. History of hypersensitivity reaction to the main ingredient of the investigational drugs
17. Patient who has administrated other drugs except donepezil for dementia treatment (it is possible to enroll after washout for 28 days)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognition Korean version(ADAS-cog) | 6 months

SECONDARY OUTCOMES:
Clinical Dementia Rating Sum of Box Korean version(CDR-SB) | 6 months
Neuropsychiatric Inventory-Q Korean version(NPI-Q) | 6 months
K-MMSE | 6 months
  Korean Mini-Mental State Examination
Korean Instrumental Activity of Daily Living(K-IADL) | 6 months
Korean Trial Masking Test-elderly's version(K-TMT-e) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Seol Heui Han, M.D., Ph.D, Principal Investigator — Konkuk University Hospital
Locations (16):
- South Korea (16):
  - The Catholic University of Korea, Bucheon, ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju-si, Jeollanam-do
  - Dong-A University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Daejeon Eulji Medical Center, Daejeon
  - Hanyang University Guri Hospital, Guri-si
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chung-ang University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No